CLINICAL TRIAL: NCT03191955
Title: Biochemical and Functional Biomarkers of Cachexia in Cancer Patients
Brief Title: Muscle Wasting in Cancer (MWIC)
Acronym: MWIC
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: Surg2015MWIC
Record Dates: First submitted 2017-05-30; First posted 2017-06-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectus Muscle Quadriceps Femoris Muscle Tumour Subcutaneous fat Intra-abdominal fat Blood Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer: Patients with oesophagogastric, hepatobiliary, and colorectal cancer for resectional surgery
- Non-cancer: Patients undergoing abdominal operation for non-inflammatory, non-cancer conditions

SUMMARY:
One way cancer affects people is through weight loss. During this weight loss (called cachexia), all types of body tissue are lost, but there is a greater rate of muscle loss than fat. Cancer patients with cachexia show decreased quality of life, decreased response to treatment (e.g. chemotherapy), increased complications from surgery, and shorter overall survival. The Investigators aim to identify molecular (and patient) factors within the tissues and bodily fluids of patients with cancer and cachexia in order to identify patients at risk of weight loss, and identify potential therapies. For this, the Investigators aim to take patient samples (muscle, fat, tumour, urine and blood) whilst patients are asleep (general anaesthesia) during their operation to remove the cancer. These samples, and similar samples taken in previous studies, will be analysed in the laboratory. Along with the sample taking, the Investigators aim to perform nutritional assessments of patients before and after surgery to get an accurate picture of their weight loss. This will include simple measurements (e.g. height/weight), and computer reanalysis of their initial diagnostic computed tomography (CT) scans (this study will not require any additional scans for patients). The Investigators also aim to assess how their muscles function, by asking them to perform walk tests and wear a physical activity meter, and assess their quality of life through questionnaires. The Investigators aim to perform nutritional and functional assessments pre-surgery and at 2-3 appointments post-surgery, up to a period of 12 months. At these timepoints, the Investigators also aim to take repeat blood and urine samples, and where possible, one additional thigh muscle biopsy. Repeated assessments allow comparison between "cancer" and "cured" states. The study will take 2 years for patient recruitment.

For comparison, the Investigators also aim to examine similar tissue and fluid samples (except tumour) from non-cancer patients who are having surgery for benign conditions (e.g. hernia).

DETAILED DESCRIPTION:
Patients: Patients with upper and lower gastrointestinal cancer for planned resectional surgery will be recruited. Patients will be identified by the clinical team at the relevant multidisciplinary team meeting and then approached for study information and consent in the surgical clinic. Age-matched, healthy controls undergoing elective surgery for benign conditions (e.g. hernias) will also be recruited.

Patient Phenotyping: CT scans performed as a routine part of diagnosis and staging will be used for analysis of body composition. All patients recruited will have their CT scans analysed where present. Control patients (e.g. hernias) may not have CT scans, but where available, will be analysed. A transverse CT image from the third lumbar vertebrae will be assessed and tissue volumes estimated by a single trained observer. Cross-sectional area for muscle and adipose tissue will be normalized for stature (cm2/m2). Estimates of whole body stores will be generated from raw data (cm2) using regression equations. Cutoffs for low muscularity are based on CT-based sarcopenia plus obesity studies of cancer patients. In a previous study, the median time to muscle biopsy after CT scan was 18 days. Phenotyping will also involve measuring basic physical attributes (e. g. weight, height etc) and self-reported physical abilities (through questionnaires).

Muscle function/Physical activity assessment: An objective assessment of physical ability will be undertaken in the clinic for all patients. This will involve a "timed up and go" test and a "6 minute walk" test. These tests have been well-validated in the literature and have good inter-rater reliability. Whilst they do add a slight burden of inconvenience to the patient clinic visit this is minimal. Additionally, a physical activity meter will be applied to the patients' thigh under a waterproof dressing. The Investigators have validated these meters in cancer patients, and they are small (35x53x7mm) and light (20g). When used in previous studies as above the patients have found them unobtrusive and they have been well-tolerated. Where possible, the Investigators will ask the patients to repeat the "timed up and go" and "6 minute walk test" in postoperative clinic up to 12 months after surgery.

Patient self-reported assessment: At routine clinic, all patients will be asked to complete validated questionnaires regarding their physical health, and their perceptions of this. These will be used to assess severity of co-morbidity, and also to assess frailty. Example questionnaires include the Scottish Co-Morbidity Severity Score, the Charlson Co-morbidity Index, and the Edmonton Frail Scale. Other questionnaires relating to self-reported appetite and function will be considered but the overall aim will be to ask select questions to reduce the burden of questioning and prevent questionnaire fatigue. The Investigators will ask participants to repeat these questionnaires in routine clinic up to 12 months post surgery.

Blood and urine sampling: At routine National Health Service (NHS) clinic, all patients will be asked to provide a blood and a urine sample. Where this is not possible, the research team will ask for permission to take these samples under general anaesthetic at planned surgery via urinary and vascular catheters inserted as part of routine care. In the postoperative phase the Investigators will ask participants to provide blood and urine samples, where possible, in routine clinic up to 12 months following surgery.

Muscle Biopsy: A biopsy of rectus abdominis muscle will be taken at surgery by the operating surgeon for all patients. This will be taken from the incision performed for the planned surgery and requires no further incisions. Where possible, an additional needle biopsy of quadriceps (thigh muscle) will also be sampled for comparison. Samples will be cleaned of fats, blood/fibrous tissue, snap frozen in liquid nitrogen and stored at -80°C, For immunohistochemistry (IHC), muscle specimens will be stitched onto a cork, treated with optimum cutting temperature (OCT) and then lowered into cooled isopentane solvent (-190°C) prior to storage at -80°C.

Fat biopsy: A biopsy of subcutaneous fat, and where possible, visceral fat will be collected at the time of surgery for all patients by the operating surgeon. This procedure does not require any additional incisions. These samples will be snap frozen in liquid nitrogen and stored at -80°C.

Tumour biopsy: For the cancer patients, once the resection specimen has been removed at surgery, this will be taken fresh to the pathology lab where the duty pathologist will retrieve sections of tumour. This will be done without compromising clinical staging and in accordance with current procedures. The tumour samples will be divided into aliquots and snap frozen in liquid nitrogen at -80°C. This will not apply to the control group.

Repeat sampling: At follow-up NHS clinic, all patients will be asked to provide repeat blood and urine samples which will be divided into aliquots and snap frozen in liquid nitrogen at -80°C. Where the patient is amenable, they will also be asked to provide a single repeat needle biopsy of the quadriceps muscle. This will be performed in clinic under local anaesthetic using standard aseptic technique. There is some discomfort associated with the injection of local anaesthetic but this is transitory. There is also some discomfort associated with the muscle biopsy but this is short-lived and in the past has been well-tolerated. Quadriceps biopsy will be requested at routine follow-up (at around 6-8 months after surgery) only. Where possible, repeat blood and urine samples will be requested at subsequent routine follow-up appointments for the duration of the study. The Investigators would anticipate this to take place for up to 12 months postoperatively.

Immunohistochemistry (IHC) and Western Blots: These will be performed as per previous publications. For IHC, frozen muscle sections will be co-stained for laminin and myosin heavy chain or lla to distinguish fibre type. Paraffin sections may also be used and stained. The distribution of fibre types, cross-sectional area of individual fibres, and the distribution of nuclei (central versus peripheral location to assess level of regeneration) will be assessed by a proprietary image analysis platform. Potential markers for measurement will include pathways members of autophagy (beclin, lamp, anti-thymocyte globulin (ATG)); apoptosis (poly adenosine di-phosphate ribose polymerase (PARP), caspase-3); oxidative stress (nitrosylated 4-Hydroxynonenal (HNE) and ubiquitinated [K48, K63] proteins); cell stress (Nuclear factor (erythroid derived 2)-like 2 Kelch-like erythroid cell-derived protein with Cap 'N' Collar homology-associated protein 1 (NRF2KEAP1), Heat Shock Protein (HSP), endoplasmic reticulum (ER)-stress); inflammation (IkB kinase (IKK), nuclear factor kappa-light-chain-enhancer of activated B cells (NFkB)-9p65, p.38, extracellular signal-related kinase (erk)1/2, c-Jun N-terminal kinase (jnk)); satellite cell maturation (Paired Box (Pax)3, Pax7, Myogenic factor (MYF)5, M-cadherin); myogenesis (myogenin, desmin); sma/mothers against decapentaplegic(SMAD) (SMAD3, phosphoSMAD3); and P-selectin.

C - reactive protein (CRP) Analysis: Systemic inflammation (SI) will be assessed using plasma CRP concentration, which will be measured with an automated immunoturbidimetric assay by the Department of Clinical Chemistry, Royal Infirmary of Edinburgh (RIE).

These analyses will be carried out both in the University of Edinburgh and at the premises of international collaborators. Any tissue transferred out of the care of the University will be fully anonymised using unique study identifiers.

This current study is a continuation of a previous study funded and supported by Cancer Research United Kingdom (UK). As part of that study tissue samples were collected, some of which remain in the University. The Investigators intend to use these remaining samples to add power to the new samples the Investigators collect by increasing the cohort size and thus the likelihood of any potential biomarker identified being significant rather than erroneous. In addition, including these samples in the analysis will add to their value, over and above that already gained by inclusion in the previous project.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified at multidisciplinary team meetings (MDT) as having oesophagogastric, hepatobiliary, and colorectal cancer suitable for resection
* Patients over 18 years of age
* Patients identified at surgical clinic as being planned for an abdominal operation for a non-cancer, non-inflammatory condition

Exclusion Criteria:

* Patients with inflammatory conditions or other condition other than cancer that might cause muscle wasting
* Patients without the capacity to consent
* Members of vulnerable groups
* Patients not undergoing abdominal surgery
* Patients undergoing totally minimally invasive (laparoscopic) surgery, with no open or hand-assisted component affording easy access to rectus muscle biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the NHS Lothian oesophagogastric, hepatobiliary, and colorectal MDT will be screened for eligibility. In addition, patients attending NHS Lothian outpatient clinics will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle index of cancer and control patients | Analysis of CT scans performed between diagnosis and operation, up to 16 weeks from diagnosis
  CT measured muscularity performed on preoperative CT scans using validated software

SECONDARY OUTCOMES:
Biochemical analysis of rectus muscle biopsies | Performed in batches on rectus biopsies taken at time of operation, within 6 months of operation
  The soluble protein content of Rectus muscle, as measured by the bicinchoninic acid assay (BCA) method.
Cancer patient 5-year postoperative survival | Up to 5 years postoperatively
  Time between operative intervention and patient death as recorded in clinical record
Measurement of patients BMI | Performed at clinic between diagnosis and operation, up to 16 weeks from date of diagnosis
  Height and weight will be measured and combined to report BMI in kg/m^2
Detailed phenotyping of patients gait speed | Performed at preoperative clinic, up to 16 weeks from date of diagnosis
  Gait speed will be measured over a defined distance to produce a gait speed in metres per second
Detailed description of patients quality of life | Performed at clinic before operation, up to 16 weeks from date of diagnosis
  Quality of life will be measured using the "QLQ-C30" questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Ramage, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data (IPD), including phenotypic data but not including patient identifiable data will be shared with other researchers in collaboration with our research group. Interested parties may contact the lead researcher with data requests.

REFERENCES:
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Background] MacDonald AJ, Greig CA, Baracos V. The advantages and limitations of cross-sectional body composition analysis. Curr Opin Support Palliat Care. 2011 Dec;5(4):342-9. doi: 10.1097/SPC.0b013e32834c49eb. PMID 21986910
- [Background] Awad S, Tan BH, Cui H, Bhalla A, Fearon KC, Parsons SL, Catton JA, Lobo DN. Marked changes in body composition following neoadjuvant chemotherapy for oesophagogastric cancer. Clin Nutr. 2012 Feb;31(1):74-7. doi: 10.1016/j.clnu.2011.08.008. Epub 2011 Aug 27. PMID 21875767
- [Background] Khal J, Hine AV, Fearon KC, Dejong CH, Tisdale MJ. Increased expression of proteasome subunits in skeletal muscle of cancer patients with weight loss. Int J Biochem Cell Biol. 2005 Oct;37(10):2196-206. doi: 10.1016/j.biocel.2004.10.017. Epub 2004 Dec 7. PMID 16125116
- [Background] Eley HL, Skipworth RJ, Deans DA, Fearon KC, Tisdale MJ. Increased expression of phosphorylated forms of RNA-dependent protein kinase and eukaryotic initiation factor 2alpha may signal skeletal muscle atrophy in weight-losing cancer patients. Br J Cancer. 2008 Jan 29;98(2):443-9. doi: 10.1038/sj.bjc.6604150. Epub 2007 Dec 18. PMID 18087277
- [Background] Stephens NA, Gallagher IJ, Rooyackers O, Skipworth RJ, Tan BH, Marstrand T, Ross JA, Guttridge DC, Lundell L, Fearon KC, Timmons JA. Using transcriptomics to identify and validate novel biomarkers of human skeletal muscle cancer cachexia. Genome Med. 2010 Jan 15;2(1):1. doi: 10.1186/gm122. PMID 20193046
- [Background] Johns N, Stephens NA, Preston T. Muscle protein kinetics in cancer cachexia. Curr Opin Support Palliat Care. 2012 Dec;6(4):417-23. doi: 10.1097/SPC.0b013e328359e6dd. PMID 23123817
- [Background] Johns N, Stephens NA, Fearon KC. Muscle wasting in cancer. Int J Biochem Cell Biol. 2013 Oct;45(10):2215-29. doi: 10.1016/j.biocel.2013.05.032. Epub 2013 Jun 11. PMID 23770121
- [Background] Skipworth RJ, Stewart GD, Bhana M, Christie J, Sturgeon CM, Guttridge DC, Cronshaw AD, Fearon KC, Ross JA. Mass spectrometric detection of candidate protein biomarkers of cancer cachexia in human urine. Int J Oncol. 2010 Apr;36(4):973-82. doi: 10.3892/ijo_00000577. PMID 20198343
- [Background] Stephens NA, Skipworth RJ, Fearon KC. Cachexia, survival and the acute phase response. Curr Opin Support Palliat Care. 2008 Dec;2(4):267-74. doi: 10.1097/SPC.0b013e3283186be2. PMID 19060563
- [Background] Tan BH, Fladvad T, Braun TP, Vigano A, Strasser F, Deans DA, Skipworth RJ, Solheim TS, Damaraju S, Ross JA, Kaasa S, Marks DL, Baracos VE, Skorpen F, Fearon KC; European Palliative Care Research Collaborative. P-selectin genotype is associated with the development of cancer cachexia. EMBO Mol Med. 2012 Jun;4(6):462-71. doi: 10.1002/emmm.201200231. Epub 2012 Apr 4. PMID 22473907
- [Background] Brzeszczynska J, Johns N, Schilb A, Degen S, Degen M, Langen R, Schols A, Glass DJ, Roubenoff R, Greig CA, Jacobi C, Fearon KCh, Ross JA. Loss of oxidative defense and potential blockade of satellite cell maturation in the skeletal muscle of patients with cancer but not in the healthy elderly. Aging (Albany NY). 2016 Aug;8(8):1690-702. doi: 10.18632/aging.101006. PMID 27454226
- [Background] Fearon KC. Cancer cachexia and fat-muscle physiology. N Engl J Med. 2011 Aug 11;365(6):565-7. doi: 10.1056/NEJMcibr1106880. No abstract available. PMID 21830971
- [Background] Das SK, Eder S, Schauer S, Diwoky C, Temmel H, Guertl B, Gorkiewicz G, Tamilarasan KP, Kumari P, Trauner M, Zimmermann R, Vesely P, Haemmerle G, Zechner R, Hoefler G. Adipose triglyceride lipase contributes to cancer-associated cachexia. Science. 2011 Jul 8;333(6039):233-8. doi: 10.1126/science.1198973. Epub 2011 Jun 16. PMID 21680814
- [Background] Mracek T, Stephens NA, Gao D, Bao Y, Ross JA, Ryden M, Arner P, Trayhurn P, Fearon KC, Bing C. Enhanced ZAG production by subcutaneous adipose tissue is linked to weight loss in gastrointestinal cancer patients. Br J Cancer. 2011 Feb 1;104(3):441-7. doi: 10.1038/sj.bjc.6606083. Epub 2011 Jan 18. PMID 21245862
- [Background] Skipworth RJ, Husi H, Ross JA. How close are we to finding noninvasive markers for upper GI tract cancer? Future Oncol. 2011 Oct;7(10):1121-4. doi: 10.2217/fon.11.90. No abstract available. PMID 21992724
- [Background] Husi H, Barr JB, Skipworth RJ, Stephens NA, Greig CA, Wackerhage H, Barron R, Fearon KC, Ross JA. The Human Urinary Proteome Fingerprint Database UPdb. Int J Proteomics. 2013;2013:760208. doi: 10.1155/2013/760208. Epub 2013 Oct 9. PMID 24222850
- [Background] Husi H, Skipworth RJ, Cronshaw A, Stephens NA, Wackerhage H, Greig C, Fearon KC, Ross JA. Programmed cell death 6 interacting protein (PDCD6IP) and Rabenosyn-5 (ZFYVE20) are potential urinary biomarkers for upper gastrointestinal cancer. Proteomics Clin Appl. 2015 Jun;9(5-6):586-96. doi: 10.1002/prca.201400111. Epub 2015 May 8. PMID 25644331
- [Background] Deans DA, Tan BH, Wigmore SJ, Ross JA, de Beaux AC, Paterson-Brown S, Fearon KC. The influence of systemic inflammation, dietary intake and stage of disease on rate of weight loss in patients with gastro-oesophageal cancer. Br J Cancer. 2009 Jan 13;100(1):63-9. doi: 10.1038/sj.bjc.6604828. PMID 19127266
- [Background] Deans DA, Wigmore SJ, Gilmour H, Paterson-Brown S, Ross JA, Fearon KC. Elevated tumour interleukin-1beta is associated with systemic inflammation: A marker of reduced survival in gastro-oesophageal cancer. Br J Cancer. 2006 Dec 4;95(11):1568-75. doi: 10.1038/sj.bjc.6603446. Epub 2006 Nov 7. PMID 17088911
- [Background] Deans DA, Tan BH, Ross JA, Rose-Zerilli M, Wigmore SJ, Howell WM, Grimble RF, Fearon KC. Cancer cachexia is associated with the IL10 -1082 gene promoter polymorphism in patients with gastroesophageal malignancy. Am J Clin Nutr. 2009 Apr;89(4):1164-72. doi: 10.3945/ajcn.2008.27025. Epub 2009 Feb 25. PMID 19244371
- [Background] Stewart GD, Skipworth RJ, Pennington CJ, Lowrie AG, Deans DA, Edwards DR, Habib FK, Riddick AC, Fearon KC, Ross JA. Variation in dermcidin expression in a range of primary human tumours and in hypoxic/oxidatively stressed human cell lines. Br J Cancer. 2008 Jul 8;99(1):126-32. doi: 10.1038/sj.bjc.6604458. PMID 18594538
- [Background] Stephens NA, Skipworth RJ, Gallagher IJ, Greig CA, Guttridge DC, Ross JA, Fearon KC. Evaluating potential biomarkers of cachexia and survival in skeletal muscle of upper gastrointestinal cancer patients. J Cachexia Sarcopenia Muscle. 2015 Mar;6(1):53-61. doi: 10.1002/jcsm.12005. Epub 2015 Mar 31. PMID 26136412
- [Background] Tan BH, Birdsell LA, Martin L, Baracos VE, Fearon KC. Sarcopenia in an overweight or obese patient is an adverse prognostic factor in pancreatic cancer. Clin Cancer Res. 2009 Nov 15;15(22):6973-9. doi: 10.1158/1078-0432.CCR-09-1525. Epub 2009 Nov 3. PMID 19887488
- [Background] Skipworth RJ, Stene GB, Dahele M, Hendry PO, Small AC, Blum D, Kaasa S, Trottenberg P, Radbruch L, Strasser F, Preston T, Fearon KC, Helbostad JL; European Palliative Care Research Collaborative (EPCRC). Patient-focused endpoints in advanced cancer: criterion-based validation of accelerometer-based activity monitoring. Clin Nutr. 2011 Dec;30(6):812-21. doi: 10.1016/j.clnu.2011.05.010. Epub 2011 Jul 5. PMID 21733604
- [Background] Grose D, Morrison DS, Devereux G, Jones R, Sharma D, Selby C, Docherty K, McIntosh D, Louden G, Nicolson M, McMillan DC, Milroy R; Scottish Lung Cancer Forum. Comorbidities in lung cancer: prevalence, severity and links with socioeconomic status and treatment. Postgrad Med J. 2014 Jun;90(1064):305-10. doi: 10.1136/postgradmedj-2013-132186. Epub 2014 Mar 27. PMID 24676985
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Rolfson DB, Majumdar SR, Tsuyuki RT, Tahir A, Rockwood K. Validity and reliability of the Edmonton Frail Scale. Age Ageing. 2006 Sep;35(5):526-9. doi: 10.1093/ageing/afl041. Epub 2006 Jun 6. No abstract available. PMID 16757522
- [Background] Trappe TA, Lindquist DM, Carrithers JA. Muscle-specific atrophy of the quadriceps femoris with aging. J Appl Physiol (1985). 2001 Jun;90(6):2070-4. doi: 10.1152/jappl.2001.90.6.2070. PMID 11356767
- [Background] Fearon KC, Preston T. Body composition in cancer cachexia. Infusionstherapie. 1990 Apr;17 Suppl 3:63-6. doi: 10.1159/000222558. No abstract available. PMID 2169464
- [Background] Acharyya S, Butchbach ME, Sahenk Z, Wang H, Saji M, Carathers M, Ringel MD, Skipworth RJ, Fearon KC, Hollingsworth MA, Muscarella P, Burghes AH, Rafael-Fortney JA, Guttridge DC. Dystrophin glycoprotein complex dysfunction: a regulatory link between muscular dystrophy and cancer cachexia. Cancer Cell. 2005 Nov;8(5):421-32. doi: 10.1016/j.ccr.2005.10.004. PMID 16286249